CLINICAL TRIAL: NCT01659411
Title: Adult Congenital Heart Disease Quality Enhancement Research Initiative
Brief Title: Adult Congenital Heart Disease Registry (QuERI)
Status: Completed | Type: Observational
Sponsor: Actelion (Industry)
Collaborators: Canadian Heart Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: AC-052-433; CHRC2011-ACHD001 (Other: Canadian Identifier)
Record Dates: First submitted 2012-07-12; First posted 2012-08-07 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Congenital Heart Disease; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Heart Defects, Congenital | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult CHD Patients: observational
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Yearly clinical visits

SUMMARY:
Multi-center, observational, U.S.-based longitudinal program. Data will be collected prospectively for 3 years. Individual physician feedback will be provided on data collected with the purpose of improving the management of patients - quality enhancement research initiative (QuERI) process from adult patients enrolled with a history of repaired Congenital Heart Disease (CHD).

DETAILED DESCRIPTION:
Approximately 800 male and female adult patients with a history of repaired CHD will be recruited from approximately 100 cardiology practices and will be followed up every twelve months for the period of three years. Consecutive patients in each practice meeting inclusion and exclusion criteria should be considered for the study. Two groups of subjects will be enrolled based on identical exclusion criteria and inclusion criteria, with the exception only of inclusion criteria #3: cohort 1- those demonstrating historic high risk criteria and cohort 2 - those demonstrating current high risk criteria.

ELIGIBILITY:
Inclusion Criteria: Cohort 1 (historic high risk)

1. Male and female adults (≥ 18 years of age)
2. Patients with documented history (at least one year) of an isolated, repaired congenital heart defect such as ASD, VSD, PDA, AVC (AVSD)
3. History of a large defect prior to closure as evidenced by any one of the following:

   * Size of: ASD > 2 cm; VSD > 1 cm; PDA > 0.6 cm
   * Shunt 2:1 or greater
   * Pre-operative PH (PAS > 40 mmHg) or documented shunt- related heart failure (radiographic evidence)
   * Pre-operative atrial fibrillation or flutter
4. High risk features (any one the following):

   * Age > 40 years
   * Later surgical repair:

     i. ≥ 2 years of age for PDA or VSD ii. ≥ 1 year of age for AVC iii. ≥ 10 years of age for ASD
   * Sinus venosus defect
   * Primum defect
   * WHO functional class > 1
   * Atrial fibrillation or flutter
5. Echocardiographic evidence of high risk features. Any one of the following:

   * Degree of TR that is mild or greater
   * Right ventricular (RV) systolic dysfunction
   * Evidence of RV dilatation: Any one of the following:

     i. Evidence of RV dilation by general, qualitative assessment ii. RV end diastolic diameter > 3.2 cm on apical 4 chamber view at the tips of the tricuspid valve iii. RV to LV ratio at end-diastole > 0.6 (RV and LV end diastolic dimensions measured from apical 4 chamber view, 1 cm apical of the respective valve annuli)
   * Any abnormality in the motion of the inter-ventricular septum
6. Ability and desire to execute the consent for follow up

Inclusion Criteria: Cohort 2 (current high risk)

1. Male and female adults (≥ 18 years of age)
2. Patients with documented history (at least one year) of an isolated, repaired congenital heart defect such as ASD, VSD, PDA, AVC (AVSD)
3. Current (within the last 12 months) evidence of 1 or more of the 7 following criteria:

   * Desaturation on exercise (92% or less)
   * 6 MWD <380 m
   * PFT demonstrating DLC <70% predicted & FEV1>70% predicted
   * ECG demonstrating i) RAD and ii) RVH or RAE
   * Physical findings of edema accompanied by elevated JVP and +HJR
   * CXR evidence of enlarged main and/or hilar pulmonary arterial shadows in association with right ventricular enlargement
   * Elevated biomarks (BNP or NT-proBNP above upper limit of normal)
4. High risk features (any one of the following:)

   * Age > 40 years
   * Later surgical repair:

     i. ≥ 2 years of age for PDA or VSD ii. ≥ 1 year of age for AVC iii. ≥ 10 years of age for ASD
   * Sinus venosus defect
   * Primum defect
   * WHO functional class > 1
   * Atrial fibrillation or flutter
5. Echocardiographic evidence of high risk features. Any one of the following:

   * Degree of TR that is mild or greater
   * Right ventricular (RV) systolic dysfunction
   * Evidence of RV dilatation: Any one of the following:

     i. Evidence of RV dilation by general, qualitative assessment ii. RV end diastolic diameter > 3.2 cm on apical 4 chamber view at the tips of the tricuspid valve iii. RV to LV ratio at end-diastole > 0.6 (RV and LV end diastolic dimensions measured from apical 4 chamber view, 1 cm apical of the respective valve annuli)
   * Any abnormality in the motion of the inter-ventricular septum
6. Ability and desire to execute the consent for follow up

Exclusion Criteria:

1. Poor mental function, drug or substance (e.g., alcohol) abuse, or unstable psychiatric illness, which, in the opinion of the investigator, may interfere with optimal participation in the study
2. Diagnosis of PAH (defined as RHC demonstrating mPAP ≥ 25 mm Hg and PCWP ≤ 15 and PVR > 3 WU or PVR (indexed) > 4 WU or treatment with PAH specific therapy) after surgical repair and prior to visit 1
3. Prior inclusion in this registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult CHD patients meeting inclusion and exclusion criteria may be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
To characterize the clinical course in a cohort of adult patients with repaired CHD at risk for developing PAH | screening (visit 1) through end of study (3 years)
  outcome measure: clinical outcomes: Assessment of function status, medications, and laboratory results, as well as an evaluation of medical history, physical examination, ECG, and echocardiography, in adult congenital heart disease patients at risk for pulmonary hypertension.

SECONDARY OUTCOMES:
To characterize the clinical outcomes in a cohort of adult patients with repaired CHD at risk for developing PAH | screening (visit 1) through end of study (3 years)
  outcome measure: clinical rate: To assess the rate of newly diagnosed pulmonary arterial hypertension in a cohort of adults with repaired congenital heart disease at risk for pulmonary arterial hypertension. To also compare clinical outcomes in patients who do and do not meet prespecified echocardiography criteria for suspected pulmonary arterial hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Landzberg, MD, Study Chair — Harvard Medical School / Boston Adult Congenital Heart

REFERENCES:
- [Derived] Landzberg MJ, Daniels CJ, Forfia P, McLaughlin VV, Bell Lynum KS, Selej M, Opotowsky AR. Timely PAH Identification in Adults With Repaired Congenital Heart Disease? The ACHD-QuERI Registry Insights. JACC Adv. 2023 Oct 31;2(9):100649. doi: 10.1016/j.jacadv.2023.100649. eCollection 2023 Nov. PMID 38938704